CLINICAL TRIAL: NCT06370325
Title: Neuromuscular Electrical Stimulation in Foot and Ankle Surgery: A Pilot Study
Brief Title: Neuromuscular Electrical Stimulation in Foot and Ankle Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00987
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the intervention group will undergo neuromuscular electrical stimulation (NMES) five days a week beginning three weeks postoperative and lasting for ten weeks. The intervention group will begin standard physical therapy at six weeks postoperative.
  Interventions: Procedure: VPOD Wireless Tens Unit; Procedure: Physical Therapy; Device: Biodex
- Control Group (Active Comparator): Participants randomized to the control group will begin standard physical therapy at six weeks postoperative.
  Interventions: Procedure: Physical Therapy; Device: Biodex

INTERVENTIONS:
Procedure: VPOD Wireless Tens Unit — The VPOD unit will deliver NMES to participants in the Intervention Group.
  Arms: Intervention Group
Procedure: Physical Therapy — Physical therapy as per standard of care.
Device: Biodex — Used to assess strength, endurance, power, and range of motion.

SUMMARY:
This is a pilot randomized controlled trial, wherein the intervention group will undergo NMES five days a week beginning three weeks postoperative and lasting for ten weeks. Both the control and intervention groups will start standard physical therapy six weeks postoperative. Primary outcome measure will be the isometric strength of the gastrocnemius muscle. The secondary outcomes will comprise subjective clinical evaluations (using the Lower Extremity Functional Scale [LEFS]), functional assessments such as the sit-to-stand test, 2-minute walk test, stair climb test and objective clinical evaluation using contralateral comparison of calf circumference.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide informed consent
* Undergoing a procedure that involves repairing an ankle fracture.

Exclusion Criteria:

Patients with medical histories that include:

* Rheumatoid arthritis
* Connective tissue disorders
* Chronic corticosteroid use
* Implanted electrical devices
* Neurological disorders
* Non-ambulatory status
* Recent surgery (within the last 3 months) that is not related to the study
* Scheduled to undergo surgery in the near future
* Epilepsy
* Diagnosed with cancer
* Have suffered acute trauma or recently have had a surgical procedure (not related to the study)
* Have cardiac problems or cardiac disease
* Have an abdominal hernia
* Have venous thrombosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Isometric Strength of Gastrocnemius Muscle | Week 6
  Measured using Biodex dynamometer.
Isometric Strength of Gastrocnemius Muscle | Week 9
  Measured using Biodex dynamometer.
Isometric Strength of Gastrocnemius Muscle | Week 12
  Measured using Biodex dynamometer.
Bilateral Calf Circumference | Week 6
Bilateral Calf Circumference | Week 9
Bilateral Calf Circumference | Week 12

SECONDARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) Questionnaire Score | Week 6
  LEFS is a 20-item questionnaire assessing functional impairment in patients with disorders affecting one or both lower extremities. Each item is rated on a scale ranging from 0 to 4: 0 indicates inability to perform the activity or extreme difficulty, 1 indicates considerable difficulty, 2 indicates moderate difficulty, 3 indicates slight difficulty, and 4 indicates no difficulty. The score is the sum of responses and ranges from a minimum of 0 to a maximum of 80, with lower scores indicating greater disability.
Lower Extremity Functional Scale (LEFS) Questionnaire Score | Week 9
  LEFS is a 20-item questionnaire assessing functional impairment in patients with disorders affecting one or both lower extremities. Each item is rated on a scale ranging from 0 to 4: 0 indicates inability to perform the activity or extreme difficulty, 1 indicates considerable difficulty, 2 indicates moderate difficulty, 3 indicates slight difficulty, and 4 indicates no difficulty. The score is the sum of responses and ranges from a minimum of 0 to a maximum of 80, with lower scores indicating greater disability.
Lower Extremity Functional Scale (LEFS) Questionnaire Score | Week 12
  LEFS is a 20-item questionnaire assessing functional impairment in patients with disorders affecting one or both lower extremities. Each item is rated on a scale ranging from 0 to 4: 0 indicates inability to perform the activity or extreme difficulty, 1 indicates considerable difficulty, 2 indicates moderate difficulty, 3 indicates slight difficulty, and 4 indicates no difficulty. The score is the sum of responses and ranges from a minimum of 0 to a maximum of 80, with lower scores indicating greater disability.
Sit-to-Stand Test | Week 6
  The sit-to-stand test involves recording the number of stands a person can complete in 30 seconds.
Sit-to-Stand Test | Week 9
  The sit-to-stand test involves recording the number of stands a person can complete in 30 seconds.
Sit-to-Stand Test | Week 12
  The sit-to-stand test involves recording the number of stands a person can complete in 30 seconds.
2 Minute Walk Test | Week 6
  In this activity, the participant is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured
2 Minute Walk Test | Week 9
  In this activity, the participant is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured
2 Minute Walk Test | Week 12
  In this activity, the participant is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured
Stair Climb Test | Week 6
  The stair climb test measures the amount of time a person ascends and descends a flight of stairs, while walking as quickly as they feel safe and comfortable to move.
Stair Climb Test | Week 9
  The stair climb test measures the amount of time a person ascends and descends a flight of stairs, while walking as quickly as they feel safe and comfortable to move.
Stair Climb Test | Week 12
  The stair climb test measures the amount of time a person ascends and descends a flight of stairs, while walking as quickly as they feel safe and comfortable to move.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J. Walls, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data to be used only by the research team.